CLINICAL TRIAL: NCT03812484
Title: An Evaluation of the New Jersey State Parole Board Swift, Certain, and Fair Project for Opioid-Involved High-Risk Parolees
Brief Title: An Evaluation of the NJSPB SCF Project for Opioid-Involved High-Risk Parolees
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Botec Analysis, LLC (Industry)
Responsible Party: Principal Investigator, Clarissa Manning, Director of Business Operations, Botec Analysis, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CC100
Record Dates: First submitted 2019-01-17; First posted 2019-01-23 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Substance Abuse; Criminal Behavior
MeSH Terms: conditions — Substance-Related Disorders; Criminal Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCF Parole (Experimental): Parolee supervised under the SCF Supervision model
  Interventions: Behavioral: SCF Supervision
- Parole-As-Usual (Active Comparator): Parolees are supervised under standard parole supervision practice in New Jersey.
  Interventions: Behavioral: Parole-as-Usual

INTERVENTIONS:
Behavioral: SCF Supervision — SCF Supervision entails a warning session (Orientation Hearing) where the rules of parole are laid out and parolees are told that any violation of stated parole conditions will be sanctioned with a brief jail term (typically a few days in jail). SCF Supervision includes regular random drug testing.
  Arms: SCF Parole
Behavioral: Parole-as-Usual — Parolees are supervised under standard parole supervision practice in New Jersey
  Other Names: PAU
  Arms: Parole-As-Usual

SUMMARY:
This study entails an evaluation of the New Jersey State Parole Board Swift, Certain, and Fair (SCF) Supervision Program. The purpose of the evaluation is to test whether subjects assigned to SCF Supervision perform better than those assigned to parole-as-usual (PAU).

DETAILED DESCRIPTION:
The Swift, Certain, and Fair (SCF) Supervision Program - Including Project HOPE Program provides funding to states, units of local government, territories, and federally recognized Indian tribes (as determined by the Secretary of the Interior) in an effort to enhance public safety, foster collaboration, and to improve the outcomes of individuals under the supervision of community corrections. The goals of this program are to develop and enhance SCF initiatives and implement the SCF model with fidelity, resulting in reduced recidivism and better outcomes for program participants. SCF approaches are intended to: (a) improve supervision strategies that reduce recidivism; (b) promote and increase collaboration among agencies and officials who work in community corrections and related fields to enhance swift and certain sanctions; (c) enhance the offenders' perception that the supervision decisions are fair, consistently applied, and consequences are transparent; and (d) improve the outcomes of individuals participating in these initiatives. The grantee will use awarded grant funds to support programming that provides services to up to 75 opioid involved parolees with services to divert them from a return to prison and manage underlying addictions with a combination of behavioral therapy and medication assisted treatments. The program combines sanctions with targeted reentry and treatment services.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older
* Participants must have a history of opioid use or addiction
* Participants have a history of parole violations or active parolees who are at risk for violation (this can include anyone who is reentering the active population from prison)
* Participants reside in or are moving to Ocean County; and
* Participants must have at least 6 months remaining on their Parole term

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Revocation Rate | 12 months
  Percentage of subjects in each condition who are revoked from parole and returned to prison

SECONDARY OUTCOMES:
Days Incarcerated | 12 months
  Total number of days incarcerated in jail or prison
New Charges | 12 months
  Number of new charges
Percent Positive Drug Tests | 12 months
  Percentage of random and scheduled drug tests that test positive for illicit drugs

CONTACTS AND LOCATIONS:
Overall Officials: Clarissa Manning, MPP, Principal Investigator — Botec Analysis, LLC
Locations (1):
- New Jersey Reentry Corporation, Toms River, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No